CLINICAL TRIAL: NCT06794489
Title: Longitudinal Biomarkers with Selected Outcome Measures in CMT
Acronym: CMT-BIO
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Michael W Sereda, MD, Professor of Neurology, Prof. Michael Sereda MD, University Medical Center Goettingen
Other Study IDs: 17/5/24
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: CMT1A; CMT (Charcot Marie Tooth Disease); CMT 1A; CMT - Charcot-Marie-Tooth Disease
Keywords: biomarkers; outcome measures
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and optional skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CMT patients
- Controls: Healthy age-matched controls

SUMMARY:
The goal of this study is to better understand the progression of CMT1A and identify risk factors influencing disease course. CMT1A, the most common hereditary peripheral neuropathy, shows high variability in individual phenotypes despite genetic similarity. Key objectives include analyzing determinants of phenotypic expression and documenting symptom variability over five years to capture disease dynamics.

Although incurable, novel CMT therapies are in development. Proving efficacy is challenging due to slow progression and limited sensitive outcome measures. This study aims to validate biomarkers (DNA/epigenetics and RNA/RT-PCR) and sensitive outcome measures from blood and skin of CMT patients over five years to support clinical therapy trials. Approximately 25 healthy volunteers will serve as controls, providing blood and skin samples for biomarker validation.

Additionally, the project will build a tissue collection (skin, blood, and cultured fibroblasts) from CMT patients of various subtypes for unrestricted scientific research, especially for the German CMT-NET network (NCT03386266). Scientific partners have free access to samples and data for research (commercial use is excluded). Currently, this collection includes over 100 standardized skin biopsies from CMT1A patients and is Germany's only repository for hereditary neuropathy tissue samples.

DETAILED DESCRIPTION:
Until now, only physical and electrophysiological examinations have been used to determine disease severity in patients with CMT. The CMT Neuropathy Score (CMTNS) is a valid and reliable nine-point composite scale that considers sensory and motor symptoms (Shy et al. 2005). However, its function as a severity or progression marker is controversial due to the slow deterioration over years (Wang et al. 2017). Surrogate biomarkers for disease severity and progression would serve as powerful tools for monitoring therapeutic effects in clinical studies. Currently, no practical biomarkers for CMT1A are available. A non-invasive MRI study showed changes in muscle and intramuscular fat accumulation in the lower limbs that correlated with clinical impairment (Gaeta et al. 2012). This method shows promising results as a surrogate outcome measure for clinical trials, but it is technically demanding and has so far only been tested in a small group of CMT patients and those with various other neuromuscular disorders.

Molecular analysis of body fluids or tissue samples is a promising strategy for developing clinically practical surrogate biomarkers for disease severity in CMT1A. In preliminary work by our research group, gene expression analyses of CMT rats were correlated with skin biopsies in CMT1A patients. This analysis identified several individual genes (STT2, CTSA, PPARG, CDA, ENPP1, and NRG1) that correlated with disease severity (Fledrich et al. 2017). Additional experiments using gene expression analyses of skin and the sciatic nerve (N. ischiadicus) enabled a distinction between mildly and severely affected CMT rats (Fledrich et al. 2012).

Due to the high variability in disease expression, we postulated that a large portion of disease manifestation occurs at the epigenetic level. Building on this, our initial approach revealed significant overlap between differentially methylated DNA regions and transcriptional changes in CMT rats. This finding suggested that changes in DNA methylation could contribute to altered gene expression and thus to the pathogenesis of CMT1A. Notably, two clusters contained highly upregulated transcripts enriched with genes associated with cell cycle regulation. Cell cycle regulation is linked to pmp22/gas315, the gene that causes CMT1A. Analysis of transcription factors indicated significant involvement of the important cell cycle regulator from the E2F family, along with its known downstream effector EZH2, a methylase essential for transcriptional repression in Schwann cells through methylation of histone H3.

Based on this, a recruitment of a total of 150 patients took place from 2016 to 2019, who were assessed over three visits for phenotypic variability, disease severity, and clinical scores (NCT03386266). In this translational study, rats overexpressing the Pmp22 gene and patient material were used. From 150 animals, 4 or 5 with mild and severe disease expressions, respectively, were selected. Patients were recruited through the CMT-NET network, where the CMTNSv2 was used as a disease score. RNAseq analyses identified several candidate genes that overlapped in both CMT1A patients and the rat models, indicating potential markers for disease severity.

These preliminary data provide evidence that epigenetic and other OMICs data from both CMT1A animal models and human patients can be used for bidirectional, informative translation in both forward and backward directions. Based on these bidirectional data, RNA sequencing was conducted from the blood of patients in CMT-NET, where initial potential biomarkers, disease modifiers, and surrogate markers were identified (Linhoff et al., publication in preparation). The rt-PCR data provide insights into predictive statements about patients' clinical development over time.

Based on these findings, we plan to further investigate the identified biomarkers in a 4th visit, following our latest ethics application to CMT-NET, and confirm their presence in skin biopsies. The focus is particularly on markers associated with newly observed symptoms, such as autonomic dysfunction and tremors. This expanded approach aims to improve the diagnosis and monitoring of the disease, enabling more precise and individualized therapeutic approaches.

The aim of this project is to better understand the natural progression of CMT1A disease and to identify potential risk factors that may influence the course of the disease. CMT1A, a subtype of CMT, is the most common hereditary peripheral neuropathy. Its slow, progressive disease course shows a high variability of individual phenotypes despite genetic homogeneity. The primary goal of the project is to analyze potential determinants of phenotypic expression, including severity levels, and to document symptom variability over a total period of five years as an indicator of disease dynamics.

CMT is a rare, incurable disease, though novel pharmacotherapies are currently being developed. Demonstrating efficacy in clinical trials is challenging due to the slow progression and lack of sensitive outcome measures. The main goal of this subproject is to validate identified biomarkers (DNA/epigenetics and RNA/RT-PCR) and selected sensitive outcome measures in the blood and skin of CMT patients over an observation period of at least 5 years to improve the assessment of efficacy in future clinical therapy trials, including diagnostic monitoring of disease progression in CMT patients. Approximately 25 healthy volunteers will also be included as controls. For the volunteers, a brief medical history will be recorded, and blood and skin samples will be collected to validate the biomarkers.

The goal of this subproject is to collect tissue samples (skin, blood, and cultured fibroblasts) from CMT patients with various subtypes for unrestricted scientific and medical research purposes, for example, for research projects within the German CMT-NET network. Scientific partners will receive free access to the samples and data. Commercial use outside of research purposes is not intended. With the help of the CMT tissue collection, CMT-NET partners can conduct morphological and molecular biological analyses of patient material, as well as utilize fibroblast cultures. Genotype-phenotype studies can also be conducted. To date, a collection of over 100 standardized skin biopsies from clinically well-characterized CMT1A patients already exists. This collection is the only tissue repository for tissue samples from patients with hereditary neuropathies in Germany.

The aim of this project is to better understand the natural progression of CMT1A disease and to identify potential risk factors that may influence the course of the disease. CMT1A, a subtype of CMT, is the most common hereditary peripheral neuropathy. Its slow, progressive disease course shows a high variability of individual phenotypes despite genetic homogeneity. The primary goal of the project is to analyze potential determinants of phenotypic expression, including severity levels, and to document symptom variability over a total period of five years as an indicator of disease dynamics.

CMT is a rare, incurable disease, though novel pharmacotherapies are currently being developed. Demonstrating efficacy in clinical trials is challenging due to the slow progression and lack of sensitive outcome measures. The main goal of this subproject is to validate identified biomarkers (DNA/epigenetics and RNA/RT-PCR) and selected sensitive outcome measures in the blood and skin of CMT patients over an observation period of at least 5 years to improve the assessment of efficacy in future clinical therapy trials, including diagnostic monitoring of disease progression in CMT patients. Approximately 25 healthy volunteers will also be included as controls. For the volunteers, a brief medical history will be recorded, and blood and skin samples will be collected to validate the biomarkers.

The goal of this subproject is to collect tissue samples (skin, blood, and cultured fibroblasts) from CMT patients with various subtypes for unrestricted scientific and medical research purposes, for example, for research projects within the German CMT-NET network. Scientific partners will receive free access to the samples and data. Commercial use outside of research purposes is not intended. With the help of the CMT tissue collection, CMT-NET partners can conduct morphological and molecular biological analyses of patient material, as well as utilize fibroblast cultures. Genotype-phenotype studies can also be conducted. To date, a collection of over 100 standardized skin biopsies from clinically well-characterized CMT1A patients already exists. This collection is the only tissue repository for tissue samples from patients with hereditary neuropathies in Germany.

The aim of this project is to better understand the natural progression of CMT1A disease and to identify potential risk factors that may influence the course of the disease. CMT1A, a subtype of CMT, is the most common hereditary peripheral neuropathy. Its slow, progressive disease course shows a high variability of individual phenotypes despite genetic homogeneity. The primary goal of the project is to analyze potential determinants of phenotypic expression, including severity levels, and to document symptom variability over a total period of five years as an indicator of disease dynamics.

CMT is a rare, incurable disease, though novel pharmacotherapies are currently being developed. Demonstrating efficacy in clinical trials is challenging due to the slow progression and lack of sensitive outcome measures. The main goal of this subproject is to validate identified biomarkers (DNA/epigenetics and RNA/RT-PCR) and selected sensitive outcome measures in the blood and skin of CMT patients over an observation period of at least 5 years to improve the assessment of efficacy in future clinical therapy trials, including diagnostic monitoring of disease progression in CMT patients. Approximately 25 healthy volunteers will also be included as controls. For the volunteers, a brief medical history will be recorded, and blood and skin samples will be collected to validate the biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical CMT Diagnosis / Anamnestically Healthy Control Group
* Genetic confirmation of CMT in adult patients
* Ability to achieve the outcome measure at baseline
* Age between 18 and 65 years
* Capacity of all study participants to consent and signed informed consent, including patient or participant information and consent form

Exclusion Criteria:

* Pregnancy or breastfeeding period
* Other relevant neurological or psychiatric disorders, acute or in the past history
* Presence of a serious previous internal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants from the Biomarkers and Validation of Selected Outcome Measures (CMTNSmod) study (ClinicalTrials.gov ID NCT03386266)
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-08-05 (Estimated)

PRIMARY OUTCOMES:
CMTNSv2, CMTNsv2-R | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  CMTNSv2 A validated composite scale that considers sensory and motor symptoms of both upper and lower extremities, as well as the ulnar nerve compound muscle action potential (CMAP) and sensory action potential (SAP) amplitudes. Version 2 of the CMT-NS has been newly designed to address various limitations of the original CMT-NS.
  CMTNSv2-R (Rasch) A modified version of CMTNSv2 using Rasch analysis to transform data into a linear measurement scale. This enables more accurate and precise quantification of functional limitations in CMT patients compared to the traditional CMTS.

SECONDARY OUTCOMES:
ONLS | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  The Overall Neuropathy Limitations Scale (ONLS) is an assessment scale designed to capture functional limitations and disabilities in patients with neuropathy. ONLS focuses on evaluating motor function, mobility, and the impact of neuropathy on patients' daily activities.
SF-36 | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  SF-36 (Short form-36) The SF-36 consists of 36 questions that inquire about the patient's overall health status and is validated in the German version.
FSS | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  Fatigue in adults is measured by the Fatigue Severity Scale (FSS).
PSQI | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  Sleep quality is assessed using the PSQI
ESS | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  Daytime sleepiness is evaluated in adults with the ESS (Epworth Sleepiness Scale).
6MWT | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  6-minute walk test
10MWT | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  10 meter walk test
Walk-12 | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  A questionnaire completed by patients to assess walking ability, consisting of twelve items, each with five response options.
Maximal Voluntary Isometric Contraction (MVIC) | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  Measured using a portable myometer (Citec, Groningen, NL) for the distal arm (grip strength, three-point pinch) and leg (dorsiflexion and plantarflexion of the foot using a stabilizing apparatus). Three tests are performed for each movement on the dominant side, with the best attempt recorded.
Nine-Hole Peg Test (9-HPT) | Change from baseline at the first timepoint of the CMT-NET biomarker study (NCT03386266) 2016/2019 to the end of the current study 2024/2025 (in total 8-9 years).
  The 9-HPT is a brief, standardized, quantitative test of upper extremity function. Both the dominant and non-dominant hand are tested twice. The 9-HPT score is calculated as the average of the four tests. A practice test for each side is conducted before starting the initial baseline measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided